CLINICAL TRIAL: NCT03866447
Title: Vitamin D and Its Topical Analogues: A Possible Role in the Pathogenesis and Treatment of Acne Vulgaris
Brief Title: Role of Vitamin D and Its Topical Analogues in Pathogenesis and Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ali saleh ali, Dermatology Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin D, and Acne
Record Dates: First submitted 2019-02-27; First posted 2019-03-07 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Vitamin D; Adapalene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin D versus placebo (Active Comparator): This group will be treated by topical Vitamin D analogue (Calcipotriol) versus placebo (panthenol).split face.half of the face will be treated by vitamin d and the other by placebo(panthenol)
  Interventions: Drug: Vitamin D analog
- Adapalene versus placebo (Active Comparator): this group will be treated by topical Adapalene (0.1%) versus versus placebo (panthenol).split face.half of the face will be treated by vitamin d and the other by placebo(panthenol)
  Interventions: Drug: Adapalene

INTERVENTIONS:
Drug: Vitamin D analog — Patients will be clinically and photographically evaluated at baseline and at each follow up visit every month for 3 months. Any local or systemic clinical side effects of the medications will be noted during each follow up visit.
  Arms: vitamin D versus placebo
Drug: Adapalene — Patients will be clinically and photographically evaluated at baseline and at each follow up visit every
  Arms: Adapalene versus placebo

SUMMARY:
Acne vulgaris is a chronic skin disease of the pilosebaceous unit characterized by formation of papules, pustules, comedones, nodules and cysts. It can have a major psychological burden on the patients. It develops due to blockage of the hair follicles. This is thought to occur as a result of the following four abnormal processes: a higher than normal amount of sebum production, excessive deposition of keratin leading to comedo formation, hair follicles' colonization by Propionibacterium acnes (P. acnes) and the local release of pro-inflammatory mediators. Androgens also play a role in pathogenesis either from elevated levels or exacerbated response

DETAILED DESCRIPTION:
In 2015, acne was estimated to affect 633 million people globally, making it the 8th most common disease worldwide. Acne commonly occurs in adolescence and affects an estimated 80-90% of teenagers. Children and adults may also be affected before and after puberty Many treatment options for acne are available, including lifestyle changes; such as eating healthy, medications (topical and systemic) and medical procedure.Despite of the availability of many therapeutic modalities, none of them has proved to be ideal. Recently, Vitamin D was proved to be an exciting option for treating many chronic inflammatory dermatological diseases. It appears to have systemic antimicrobial and other effects that may be crucial in a variety of both acute and chronic illnesses. Vitamin D regulates the immune system, Furthermore, it has antioxidant and anti-comedogenic properties. So, Vitamin D deficiency maybe involved in the pathogenesis of Acne Vulgaris . Thus,Vitamin D use could potentially reduce inappropriate antibiotic prescription and boost therapeutic response, either as a monotherapy or in combination with other anti-acne medications. High glycemic food intake and excessive consumption of dairy products as well as of saturated fatty acids were all suggested to have an influence on AV course. In addition, obesity has been reported to be associated with acne. Interestingly, genetic studies found out that obesity can drive down vitamin D levels So, there seems to be a theoretical background about the association between Acne Vulgaris, Vitamin D and obesity

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Acne of any grade.
2. Patients between 18 and 45 years old.

Exclusion Criteria:

1. Patients below 18 and above 45years.
2. Patients with any concomitant Dermatologic or systemic illness
3. Patients on any topical or systemic medication within 4 weeks before enrollment.
4. Pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of topical Vitamin D analogues in treatment of Acne Vulgaris. | 3 months
  patients will be evaluated before and after treatment with Vitamin D and Adapalene versus placebo(panthenol).patients with acne will be graded according to Facial Acne Severity Scale. This scale is based on half-face counting of inflammatory lesions .Mild 0-5 Moderate 6-20 Severe 21-50 Very severe >50

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slaby O, McDowell A, Bruggemann H, Raz A, Demir-Deviren S, Freemont T, Lambert P, Capoor MN. Is IL-1beta Further Evidence for the Role of Propionibacterium acnes in Degenerative Disc Disease? Lessons From the Study of the Inflammatory Skin Condition Acne Vulgaris. Front Cell Infect Microbiol. 2018 Aug 14;8:272. doi: 10.3389/fcimb.2018.00272. eCollection 2018. PMID 30155445
- [Background] Al-Taiar A, AlKhabbaz M, Rahman A, Al-Sabah R, Shaban L, Akhtar S. Plasma 25-Hydroxy Vitamin D is not Associated with Acne Vulgaris. Nutrients. 2018 Oct 17;10(10):1525. doi: 10.3390/nu10101525. PMID 30336597
- [Background] Karimkhani C, Dellavalle RP, Coffeng LE, Flohr C, Hay RJ, Langan SM, Nsoesie EO, Ferrari AJ, Erskine HE, Silverberg JI, Vos T, Naghavi M. Global Skin Disease Morbidity and Mortality: An Update From the Global Burden of Disease Study 2013. JAMA Dermatol. 2017 May 1;153(5):406-412. doi: 10.1001/jamadermatol.2016.5538. PMID 28249066
- [Background] Jia X, Liu J, Chen B, Jin D, Fu Z, Liu H, Du S, Popkin BM, Mendez MA. Differences in nutrient and energy contents of commonly consumed dishes prepared in restaurants v. at home in Hunan Province, China. Public Health Nutr. 2018 May;21(7):1307-1318. doi: 10.1017/S1368980017003779. Epub 2018 Jan 8. PMID 29306339
- [Background] Reichrath J, Zouboulis CC, Vogt T, Holick MF. Targeting the vitamin D endocrine system (VDES) for the management of inflammatory and malignant skin diseases: An historical view and outlook. Rev Endocr Metab Disord. 2016 Sep;17(3):405-417. doi: 10.1007/s11154-016-9353-4. PMID 27447175
- [Background] Rocha MA, Bagatin E. Skin barrier and microbiome in acne. Arch Dermatol Res. 2018 Apr;310(3):181-185. doi: 10.1007/s00403-017-1795-3. Epub 2017 Nov 17. PMID 29147769
- [Background] Cooper AJ, Harris VR. Modern management of acne. Med J Aust. 2017 Jan 16;206(1):41-45. doi: 10.5694/mja16.00516. PMID 28076744
- [Background] Hayashi N, Akamatsu H, Kawashima M; Acne Study Group. Establishment of grading criteria for acne severity. J Dermatol. 2008 May;35(5):255-60. doi: 10.1111/j.1346-8138.2008.00462.x. PMID 18477223
- [Background] Aspray TJ, Bowring C, Fraser W, Gittoes N, Javaid MK, Macdonald H, Patel S, Selby P, Tanna N, Francis RM; National Osteoporosis Society. National Osteoporosis Society vitamin D guideline summary. Age Ageing. 2014 Sep;43(5):592-5. doi: 10.1093/ageing/afu093. Epub 2014 Jul 28. PMID 25074538
- [Background] Blackburn H, Jacobs D Jr. Commentary: Origins and evolution of body mass index (BMI): continuing saga. Int J Epidemiol. 2014 Jun;43(3):665-9. doi: 10.1093/ije/dyu061. Epub 2014 Apr 1. No abstract available. PMID 24691955